CLINICAL TRIAL: NCT00004937
Title: Open Label Phase II Study on XR5000 Administered as a 5 Day Infusion in Patients With Glioblastoma Multiforme
Brief Title: Acridine Carboxamide in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16991G; EORTC-16991G; XENOVA-XR5000/014/98
Record Dates: First submitted 2000-03-07; First posted 2004-08-09 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — DACA, acridine

INTERVENTIONS:
Drug: acridine carboxamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of acridine carboxamide in treating patients who have recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy acridine carboxzmide in terms of objective response rate and response duration in patients with glioblastoma multiforme. II. Determine the toxicities of this treatment regimen in this patient population.

OUTLINE: This is a multicenter study. Patients receive acridine carboxamide IV continuously over days 1-5. Treatment repeats every 3 weeks for at least 2 courses and up to a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks until disease progression.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed recurrent glioblastoma multiforme Measurable disease on contrast MRI Lesion at least 2 cm in diameter

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Karnofsky 70-100% Life expectancy: At least 3 months Hematopoietic: WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2 times ULN Transaminases no greater than 2 times ULN Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: Normal cardiac function No ischemic heart disease within the past 6 months Normal electrocardiogram Other: No unstable systemic diseases No active uncontrolled infections No prior or other concurrent malignancies except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix No psychological, familial, sociological, or geographical condition that would preclude study Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 weeks since prior adjuvant chemotherapy for brain tumor No other prior chemotherapy Endocrine therapy: Must be on stable or decreasing doses of corticosteroids for at least 2 weeks Radiotherapy: At least 3 months since prior radiotherapy to the brain No prior high dose radiotherapy No prior stereotactic boost or implant radiotherapy Surgery: No prior surgery (except biopsy) for recurrent brain tumor At least 3 months since prior surgery for primary brain tumor Other: No other concurrent anticancer agents No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Twelves, MD, BMedSci, FRCP, Study Chair — University of Glasgow
Locations (1):
- Beatson Oncology Centre, Glasgow, Scotland, United Kingdom